CLINICAL TRIAL: NCT02023528
Title: Dialysis Registry in Utah
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, University of Utah
Other Study IDs: IRB_00063655
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Based on the Medicare data, the 5-year survival of dialysis patients is only 39%. This is lower than that of stage IIIB breast cancer (54% 5-year survival). The annual mortality of dialysis patients is ~ 23% compared to <0.1% in the United States general population. Even kidney transplant recipients have a substantially higher mortality (~7%) compared to the general population. Consequently, the life-expectancy of dialysis and transplant populations is much lower than that of the general population. Cardiovascular events are the leading cause of death in dialysis patients and malnutrition is also a strong risk factor for death. The current proposal is to develop a prospective registry of incident dialysis patients at the University of Utah dialysis program to examine cardiovascular and nutritional factors in dialysis patients. This registry will include clinical and administrative data. In addition, blood samples will be stored for future analyses.

DETAILED DESCRIPTION:
Design:

This is a prospective, observational study of patients in the University of Utah dialysis program.

Study Procedures:

Patients new to dialysis at the University of Utah dialysis program will be approached to determine whether they want to participate in the registry. If they are interested, the study purpose and procedures will be explained and informed consent obtained. Participants will be asked to complete a brief questionnaire on demographics (age, gender, race, education), co-morbid conditions (diabetes mellitus, congestive heart failure, hypertension, chronic lung disease, malignancies, coronary artery disease, cerebrovascular disease and peripheral vascular disease), physical activity level, cognitive function and sleep patterns. Height, weight, and waist circumference will be measured. Annual follow up visits will be conducted with each patient until the 5th annual follow-up, death, transplantation or loss to follow-up. During these visits, participants will complete questionnaires on physical activity level, cognitive function and sleep patterns. Height, weight, and waist circumference will be measured. Thirty milliliters (ml) of blood will also be drawn.

Relevant Dialysis data (cause and duration of kidney disease, duration of dialytic therapy, duration and frequency of dialysis sessions, type of dialyzer used, type of vascular access), medications (erythropoietin dose and route of administration, iron supplements), laboratory markers (hemoglobin, serum calcium, serum intact parathyroid hormone, serum phosphorous, white blood cell count with differential neutrophil and lymphocyte counts and urea reduction rate) will be obtained from the electronic medical records.

30 ml of blood will be drawn on a dialysis day before dialysis. Serum/ plasma will be separated. DNA will be extracted from the rest of the cells in the baseline visit and stored. The samples will be stored in a freezer for future analyses.

Participants will be longitudinally followed using the dialysis unit electronic medical records and with annual follow up visits. In addition, if the participant consents, Medicare follow-up data from the United States Renal Data System (USRDS) will be obtained. The USRDS is a national registry of dialysis patients. U.S. Medicare regulations stipulate that irrespective of their insurance status, all patients starting on chronic dialysis therapy must be reported to the USRDS. The outcomes of these patients are tracked by USRDS using the Medicare database and national Vital Statistics (maintained by National Center for Health Statistics).

ELIGIBILITY:
Inclusion Criteria:

* Must be above the age of 18.
* Consenting to participate in the registry.

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New patients starting on dialysis at the University of Utah care dialysis program.
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Demographics, co-morbid conditions and characteristics of dialysis patients | baseline
  The objective is to develop a registry of incident dialysis patients at the University of Utah dialysis program

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States